CLINICAL TRIAL: NCT01535170
Title: Bovine Lactoferrin as a Natural Regimen of Selective Decontamination of the Digestive Tract in Patients With Prolonged Mechanical Ventilation
Acronym: LFasSDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Deapartment of Medical Research, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMR99-IRB-076
Record Dates: First submitted 2011-06-15; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Nosocomial Infections
Keywords: lactoferrin; selective decontamination of digestive tract; antimicrobial activity; prolonged mechanical ventilation; respiratory care center
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bovine Lactoferrin (Experimental): Lactoferrin and placebo will be masked as drug A and B in the factory. Randomization will be stratified by center and patients will be randomized into A or B groups by a random-number table sequence after informed consents are obtained. No patients, research nurses, investigators, or other medical staffs in RCC will be aware of the assignment during the study period.
  Patients will receive either bLF (10 mg/Kg/day) (Westland Co-operative Dairy Company, New Zealand) or placebo (starch) as control. The dosage of bLF is based on the mean hLF intake that very low body weight neonates ingest with mother's fresh milk in the first 2 weeks of life (30-150 mg/d) [16] and bLF 200 mg bid is found to be effective to suppress Helicobacter pylori [17]. Drug administration will begin within 24 hours after RCC admission and will last for 6 weeks or until discharge. Medication and nutritional support will be prescribed as the medical routine.
  Interventions: Dietary Supplement: bovine Lactoferrin
- Placebo (Placebo Comparator): Patients will receive either bLF (10 mg/Kg/day) (Westland Co-operative Dairy Company, New Zealand) or placebo (starch) as control.
  Interventions: Dietary Supplement: bovine Lactoferrin

INTERVENTIONS:
Dietary Supplement: bovine Lactoferrin — Patients will receive either bLF (10 mg/Kg/day) (Westland Co-operative Dairy Company, New Zealand) or placebo (starch) as control. The dosage of bLF is based on the mean hLF intake that very low body weight neonates ingest with mother's fresh milk in the first 2 weeks of life (30-150 mg/d) [16] and bLF 200 mg bid is found to be effective to suppress Helicobacter pylori [17].

SUMMARY:
Nosocomial infection with antibiotic-resistant strains is a major threat to critical care medicine. Selective decontamination of the digestive tract (SDD) is one of the strategies to reduce ventilator associated pneumonia and sepsis in critically ill patients. Lactoferrin (LF) is a natural multifunctional protein with antimicrobial, anti-tumor, antioxidant, and immunomodulatory effects. It has been shown to inhibit the growth of a number of pathogenic bacteria including antibiotic-resistant strains, fungi and even viruses in both in vitro and in vivo studies.

In a recent study, the investigators performed pathogen challenges of the digestive tract of a transgenic milk-fed animal model. The results showed that recombinant LF has broad spectrum antimicrobial activity in the digestive tract and protects the mucosa of the small intestine from injury, implying that LF can be used as an effective selective decontaminant of the digestive tract.

This study is a prospective, randomized, double-blind, placebo- controlled clinical trial examining whether oral supplementation with bLF can reduce nosocomial infection, sepsis and even mortality in patients with prolonged mechanical ventilation (MV). Patients with MV for more than 21 days and no signs of infection on admission to our Respiratory Care Center (RCC) will be enrolled. They will be randomized to receive either bovine LF (bLF, 10 mg/kg/day) or placebo for 6 weeks by center.

The primary objective is to evaluate the effectiveness of bLF in the prevention of nosocomial infection. Secondary objectives are assessment of incidence of nosocomial infection, mortality, weaning rate from MV and change of the immune system. The investigators hypothesize that bLF may 1) prevent nosocomial infection; 2) reduce mortality; 3)increase weaning rate from MV; 4)increase immunity in patients with prolonged MV.

DETAILED DESCRIPTION:
Background Nosocomial infection Nosocomial infection, especially those caused by bacteria resistant to antibiotics, is a major threat to critical care medicine. A systemic review revealed that 10-20% of patients receiving mechanical ventilation (MV) more than 48 hours will develop ventilator associated pneumonia (VAP), patients who develop VAP are twice as likely to die compared with the similar patients without VAP, and patients who develop VAP have in additional hospital costs more than $ 10,019 [1].

The same problem occurs in Respiratory Care Centers (RCCs) which are designed to care the patients with prolonged mechanical ventilation (PMV), MV for more than 21 days, in Taiwan. One report from Taiwan showed that nosocomial infection rate in RCC is about 40% and the patients develop nosocomial infection have lower weaning rate and higher mortality compared with the patients without infection [2]. It has been estimated that 50% to 60% the nosocomial infection occurring each year in the United Sates are caused by antibiotic-resistant bacterial strains [3]. This high rate of resistant strains increases the morbidity, mortality and medical costs of infection. Preventing infection and limiting the emergence of antibiotic-resistant strains are two important issues in critical care medicine.

Selective Decontamination of Digestive Tract (SDD) One of the current hypotheses of nosocomial infection is that colonization of the nasopharynx and oropharynx predisposes patients to the development of nosocomial pneumonia, and the bacterial overgrowth in the intestinal tract increases gut wall permeability, leading to bacterial translocation and sepsis. Selective decontamination of the digestive tract (SDD), which aims to eradicate colonization of potential pathogens from the oropharynx and gastrointestinal tract, is one of the strategies to reduce ventilator associated pneumonia (VAP) and sepsis in critically ill patients. Controversy exists about the effectiveness of SDD in reducing mortality and preventing antibiotic resistance [4-6]. The present SDD regimens may create selective pressure and induce the emergence of methicillin-resistant Staphylococcus aureus (MRSA), Gram-negative bacilli harboring extended-spectrum β-lactamases (ESBL), and even Candida [7, 8]. Therefore, SDD research must aim to find an ideal regimen effective on most pathogens while leaving the anaerobic flora undisturbed.

Lactoferrin Lactoferrin (LF) is an iron-binding glycoprotein found in milk and various external secretions such as saliva, tears, airway secretion, and the granules of neutrophils, implying a important role in innate immunity. This protein has a number of biological functions, including antimicrobial, anti-tumor, antioxidant, and immunomodulatory effects. Partial degradation of LF by pepsin in stomach, may give rise to peptides termed lactoferricin with more potent antimicrobial activity. LF and lactoferricin have been shown to inhibit the growth of a number of pathogenic bacteria including antibiotic-resistant strains, fungi and even viruses in both in vitro and in vivo studies [9,10]. In mouse experiments, oral administration of bovine LF reduced bacterial infections in the gastrointestinal tract [9] while promoting the growth of bacteria with low iron requirements such as Lactobacillus and Bifidobacteria, which are generally believed to be beneficial to the host [11].

Bovine lactoferrin (bLF) and human lactoferrin (hLF) have high (77%) amino acid homology, with bLF exhibiting even higher in vitro antimicrobial activity than hLF.5 Bovine lactoferrin has been granted GRAS (generally recognized as safe) status by the US Food and Drug Administration [12] and on this basis is added to infant formula by many manufacturers with no reported adverse effects. Despite many promising in vitro and animal experimental data, clinical information on bLF is scarce, with no studies investigating the effects of bLF supplementation in patients with prolonged mechanical ventilation.

Our previous studies We previously demonstrated that both recombinant porcine LF (pLF) produced from yeast [13] and a synthetic 20-residue porcine lactoferricin peptide [11] exhibit antimicrobial activity in vitro. Its bactericidal activity was four times more effective than that of human lactoferricin [14].

In our recent report [15], we performed pathogen challenges of the digestive tract of a transgenic milk-fed animal model to test if porcine LF (pLF) is an effective SDD regimen. Transgenic mice expressed recombinant LF in their milk at 120 ± 13.6 mg/L during the lactation stage and fed normal CD-1 mice pups for 4 weeks. The pups were subsequently challenged with pathogenic Escherichia coli, Staphylococcus aureus and Candida albicans. The groups that were fed pLF transgenic milk demonstrated statistically significant improvements in weight gain, lower bacterial numbers in intestinal fluid, blood and liver, and healthier microvilli in the small intestinal tissue, lower proinflammatory cytokines when compared to the control groups that were fed normal milk. Results showed that recombinant pLF expressed in the milk of transgenic mice and fed to mice pups led to broad spectrum antimicrobial activity in the digestive tract and protected the mucosa of the small intestine from injury, implying that porcine LF can be used as an effective selective decontaminant of the digestive tract.

Aim of this study This study is a prospective, randomized, double-blind, placebo-controlled clinical trial examining whether oral supplementation with bLF reduces nosocomial infection, sepsis and even mortality in patients with prolonged mechanical ventilation.

Methods Patients Between July 1, 2010, and June 30, 2012, we will enroll about 280 patients with mechanical ventilation for more than 21 days and no evident signs of infection on admission to our Respiratory Care Centers (RCCs) for clinical study. The study has been sent to the Ethics Committees of China Medical University Hospital for approval. Patients or guardians provide written informed consent after our explanation. Exclusion criteria were informed consent lacking/refused, ongoing antibiotics treatment for infection, predicted mortality in 7 days. All patients will be followed up until death or discharge from our hospital.

Objectives The primary objective is to evaluate the effectiveness of bLF in the prevention of the first episode of nosocomial infection and sepsis of bacterial or fungal origin after admission to RCC. Secondary objectives are assessments of the incidence of pneumonia, urinary tract infection and sepsis, mortality prior to discharge (overall and sepsis-attributable), weaning rate from MV, total days of MV, alteration of immune system, cytokines and liver function, and adverse effects or intolerance.

Study design Lactoferrin and placebo will be masked as drug A and B in the factory. Randomization will be stratified by center and patients will be randomized into A or B groups by a random-number table sequence after informed consents are obtained. No patients, research nurses, investigators, or other medical staffs in RCC will be aware of the assignment during the study period.

Patients will receive either bLF (10 mg/Kg/day) (Westland Co-operative Dairy Company, New Zealand) or placebo (starch) as control. The dosage of bLF is based on the mean hLF intake that very low body weight neonates ingest with mother's fresh milk in the first 2 weeks of life (30-150 mg/d) [16] and bLF 200 mg bid is found to be effective to suppress Helicobacter pylori [17]. Drug administration will begin within 24 hours after RCC admission and will last for 6 weeks or until discharge. Medication and nutritional support will be prescribed as the medical routine.

Systematic surveillance of adverse events (eg, vomiting, feeding intolerance, skin rashes) will be performed through daily examination. Weekly surveillance of liver function, complete blood counts, CD4/CD8, cytokines (TNF-alpha, IFN-gamma, IL-1, IL-2, IL-12, IL-18) will be performed [18,19].

Definition of outcomes The diagnosis of sepsis is based on the detection of clinical signs and symptoms by the physicians in charge, presence of laboratory findings consistent with sepsis, and isolation of a causative organism from blood or body fluids. Patients with an episode of sepsis continue to receive follow-up until death or discharge from RCC for secondary outcomes [16]. VAP is characterized by the presence of signs of respiratory infection (fever, leukocytosis and purulent respiratory secretions), and a new and persistent infiltrate on chest X-ray in patients undergoing MV [20]. Urinary tract infections is diagnosed by isolation of a pathogen from urine collected by suprapubic puncture or bladder catheterization, with growth of more than 100 000 bacteria/mL or more than 10 000 fungi/mL. Success of weaning from MV is defined as no need of MV for more than 5 days.

Statistical Analysis Sample size analysis predicted that a total of 131 MV patients in each group would be needed to detect a relative difference between treated and non-treated patients of at least 60% (decrease from 20% to 6%) for mortality rate based on two-sided test with type I error of 0.05 or less and 80% power of 80%. Quantitative variables will be expressed as mean and standard deviation. Categorical variables will be represented by percentages. Univariate analyses exploring associations between individual risk factors and primary/secondary outcomes were performed using Fisher's exact test for dichotomous variables and Student's t test for continuous variables. A multivariate logistic regression model is performed to investigate the effect of relevant risk factors and relative contributions of the various risk factors. Goodness of fit is evaluated through the log-likelihood of the fitted model. Odds ratios and their 95% confidence interval are calculated in the logistic regression model to describe the strength of the relationship between the categorical risk factors and outcomes. All tests are two-sided, and a p-value of 0.05 is considered to be statistically significant. All analysis is carried out using SAS software version 6.12 (SAS Institute Inc, Cary, NC).

EXPECTED FINDINGS

Our findings can be expected to answer the following questions as follows:

1. Can oral supplement of bLF prevent nosocomial infection in patients with PMV?
2. Can oral supplement of bLF reduce the incidence of nosocomial infection and reduce the use of antibiotics in patient with PMV?
3. Can oral supplement of bLF reduce mortality of the patients with PMV?
4. Can oral supplement of bLF increase the weaning rate from MV in patients with PMV?
5. What are the changes of immune system after oral supplement of bLF in patients of PMV?

EXPECTED CONTRIBUTION FROM CURRENT PROJECT Preventing infection and limiting the emergence of antibiotic-resistant strains are two important issues in critical care medicine. To find a natural antimicrobial peptide as an adjuvant therapy for antimicrobial agents in treatment of the antibiotic-resistant strains, or as a regimen to increase immunity and to prevent infection is one of the directions of researches. LF is one of the promising agents in many vitro and animal studies. The study is trying to examine if LF is an ideal natural SDD regimen for the prevention of nosocomial pneumonia or sepsis in patients with PMV. If the result is positive, LF can be used clinically to increase the survival of the critically ill patients, increase weaning rate from MV, reduce the prescription of antibiotics and finally medical cost.

REFERENCES (List without PMID No)

12. CFSAN/Office of Food Additive Safety. Agency response letter: GRAS notice No. GRN 000077. US Food and Drug Administration Web site. http:// www.fda.gov/Food/FoodIngredientsPackaging/GenerallyRecognizedasSafeGRAS/GRASListings/ucm154188.htm. August 14, 2001. Accessed May 21, 2009.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mechanical ventilation for more than 21 days and no evident signs of infection in our Respiratory Care Center (RCC).

Exclusion Criteria:

1. Informed consent lacking/refused
2. Ongoing antibiotics treatment for infection
3. Predicted mortality in 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Prevention of infection | 30 days
  To evaluate the effectiveness of bLF in the prevention of the first episode of nosocomial infection and sepsis

SECONDARY OUTCOMES:
Effects on infection | 30 days
  assessments of the incidence of pneumonia, urinary tract infection.
Effects on immunity | 30 days
  alteration of immune system, cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, China Medical Univdersity Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Background] Yen CC, Lin CY, Chong KY, Tsai TC, Shen CJ, Lin MF, Su CY, Chen HL, Chen CM. Lactoferrin as a natural regimen for selective decontamination of the digestive tract: recombinant porcine lactoferrin expressed in the milk of transgenic mice protects neonates from pathogenic challenge in the gastrointestinal tract. J Infect Dis. 2009 Feb 15;199(4):590-8. doi: 10.1086/596212. PMID 19125673
- [Background] Safdar N, Dezfulian C, Collard HR, Saint S. Clinical and economic consequences of ventilator-associated pneumonia: a systematic review. Crit Care Med. 2005 Oct;33(10):2184-93. doi: 10.1097/01.ccm.0000181731.53912.d9. PMID 16215368
- [Background] Jones RN. Resistance patterns among nosocomial pathogens: trends over the past few years. Chest. 2001 Feb;119(2 Suppl):397S-404S. doi: 10.1378/chest.119.2_suppl.397s. PMID 11171776
- [Background] de Jonge E, Schultz MJ, Spanjaard L, Bossuyt PM, Vroom MB, Dankert J, Kesecioglu J. Effects of selective decontamination of digestive tract on mortality and acquisition of resistant bacteria in intensive care: a randomised controlled trial. Lancet. 2003 Sep 27;362(9389):1011-6. doi: 10.1016/S0140-6736(03)14409-1. PMID 14522530
- [Background] Bonten MJ, Grundmann H. Selective digestive decontamination and antibiotic resistance: a balancing act. Crit Care Med. 2003 Aug;31(8):2239-40. doi: 10.1097/01.CCM.0000080491.46005.3F. No abstract available. PMID 12973186
- [Background] Pittet D, Eggimann P, Rubinovitch B. Prevention of ventilator-associated pneumonia by oral decontamination: just another SDD study? Am J Respir Crit Care Med. 2001 Aug 1;164(3):338-9. doi: 10.1164/ajrccm.164.3.2105072b. No abstract available. PMID 11500329
- [Background] Camus C, Bellissant E, Sebille V, Perrotin D, Garo B, Legras A, Renault A, Le Corre P, Donnio PY, Gacouin A, Le Tulzo Y, Thomas R. Prevention of acquired infections in intubated patients with the combination of two decontamination regimens. Crit Care Med. 2005 Feb;33(2):307-14. doi: 10.1097/01.ccm.0000152224.01949.01. PMID 15699832
- [Background] Vincent JL. Selective digestive decontamination: for everyone, everywhere? Lancet. 2003 Sep 27;362(9389):1006-7. doi: 10.1016/S0140-6736(03)14445-5. No abstract available. PMID 14522525
- [Background] Valenti P, Antonini G. Lactoferrin: an important host defence against microbial and viral attack. Cell Mol Life Sci. 2005 Nov;62(22):2576-87. doi: 10.1007/s00018-005-5372-0. PMID 16261253
- [Background] Tomita M, Wakabayashi H, Yamauchi K, Teraguchi S, Hayasawa H. Bovine lactoferrin and lactoferricin derived from milk: production and applications. Biochem Cell Biol. 2002;80(1):109-12. doi: 10.1139/o01-230. PMID 11908633
- [Background] Kim WS, Ohashi M, Tanaka T, Kumura H, Kim GY, Kwon IK, Goh JS, Shimazaki K. Growth-promoting effects of lactoferrin on L. acidophilus and Bifidobacterium spp. Biometals. 2004 Jun;17(3):279-83. doi: 10.1023/b:biom.0000027705.57430.f1. PMID 15222478
- [Background] Chen HL, Lai YW, Yen CC, Lin YY, Lu CY, Yang SH, Tsai TC, Lin YJ, Lin CW, Chen CM. Production of recombinant porcine lactoferrin exhibiting antibacterial activity in methylotrophic yeast, Pichia pastoris. J Mol Microbiol Biotechnol. 2004;8(3):141-9. doi: 10.1159/000085787. PMID 16088216
- [Background] Chen HL, Yen CC, Lu CY, Yu CH, Chen CM. Synthetic porcine lactoferricin with a 20-residue peptide exhibits antimicrobial activity against Escherichia coli, Staphylococcus aureus, and Candida albicans. J Agric Food Chem. 2006 May 3;54(9):3277-82. doi: 10.1021/jf053031s. PMID 16637685
- [Background] Manzoni P, Rinaldi M, Cattani S, Pugni L, Romeo MG, Messner H, Stolfi I, Decembrino L, Laforgia N, Vagnarelli F, Memo L, Bordignon L, Saia OS, Maule M, Gallo E, Mostert M, Magnani C, Quercia M, Bollani L, Pedicino R, Renzullo L, Betta P, Mosca F, Ferrari F, Magaldi R, Stronati M, Farina D; Italian Task Force for the Study and Prevention of Neonatal Fungal Infections, Italian Society of Neonatology. Bovine lactoferrin supplementation for prevention of late-onset sepsis in very low-birth-weight neonates: a randomized trial. JAMA. 2009 Oct 7;302(13):1421-8. doi: 10.1001/jama.2009.1403. PMID 19809023
- [Background] Okuda M, Nakazawa T, Yamauchi K, Miyashiro E, Koizumi R, Booka M, Teraguchi S, Tamura Y, Yoshikawa N, Adachi Y, Imoto I. Bovine lactoferrin is effective to suppress Helicobacter pylori colonization in the human stomach: a randomized, double-blind, placebo-controlled study. J Infect Chemother. 2005 Dec;11(6):265-9. doi: 10.1007/s10156-005-0407-x. PMID 16369731
- [Background] Mulder AM, Connellan PA, Oliver CJ, Morris CA, Stevenson LM. Bovine lactoferrin supplementation supports immune and antioxidant status in healthy human males. Nutr Res. 2008 Sep;28(9):583-9. doi: 10.1016/j.nutres.2008.05.007. PMID 19083463
- [Background] Teraguchi S, Wakabayashi H, Kuwata H, Yamauchi K, Tamura Y. Protection against infections by oral lactoferrin: evaluation in animal models. Biometals. 2004 Jun;17(3):231-4. doi: 10.1023/b:biom.0000027697.83706.32. PMID 15222470